CLINICAL TRIAL: NCT01503086
Title: Computerized Cognitive Training for Pediatric Brain Tumor Patients: A Pilot Study
Brief Title: Computer Training Program for Younger Patients With a Brain Tumor Who Underwent Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACCL10P1; NCI-2012-00112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ACCL10P1; CDR0000721387; ACCL10P1 (Other: Children's Oncology Group); COG-ACCL10P1 (Other: DCP); ACCL10P1 (Other: CTEP); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Brain Neoplasm; Recurrent Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (interactive training program) (Experimental): Patients undergo a home-based, computerized, interactive training program comprising 3-5 sessions of 15-45 minutes every week for 5-9 weeks. The program contains twelve visually engaging and interesting exercises that target skills involving visual-spatial and verbal WM. The program is adaptive in a way that each difficulty task is automatically adjusted on a trial-by-trail basis to match a patient's current WM. Each patient has an interventional coach who has online access to patient's training sessions and outcomes (pass or fail). Coaches are able to modify the training sequence or make suggestions to patients and/or parents about how progress can be maximized. Coaches also have telephone meetings with patients and/or families once a week to ensure compliance, track progress, provide feedback, and answer questions that arise during training.
  Interventions: Procedure: Cognitive Assessment; Other: Computer-Assisted Cognitive Training; Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (non-adaptive training program) (Experimental): Patients undergo a home-based, computerized, interactive, non-adaptive training program comprising 3-5 sessions of 15-45 minutes a week for 5-9 weeks. Each patient also has an interventional coach as in arm I. Patients in both arms complete a brief neuropsychological/behavioral assessment comprising the WIS-IV, the CMS, and the CVLT-C at baseline, after completion of study, and at 6 months after completion of study. Additionally, parents complete a parent-report questionnaire to gather information about patient's behaviors, thoughts, emotions, adaptive skills, and social and functional impairment. Parents and children also complete surveys about the program regarding technical feasibility, adherence, ease-of-use, and satisfaction.
  Interventions: Procedure: Cognitive Assessment; Other: Computer-Assisted Cognitive Training; Procedure: Psychosocial Assessment and Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies
Other: Computer-Assisted Cognitive Training — Receive computer-assisted cognitive training
Procedure: Psychosocial Assessment and Care — Ancillary studies
  Other Names: Psychosocial Care/Assessment
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well an adaptive computerized cognitive training program works compared to a non-adaptive computerized cognitive training program in treating younger patients with brain tumor who underwent radiation therapy. Providing a computer training program may improve the well-being and quality of life of patients with cognitive (physical and mental) function difficulties caused by radiation therapy to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of a home-based, computerized, cognitive training program for patients with pediatric brain tumors who are undergoing cranial radiation therapy (CRT), treated in multiple Children Oncology Group (COG) institutions.

EXPLORATORY OBJECTIVES:

I. To estimate the effect size of this program on measures of attention and working memory in patients with brain tumors treated with CRT in order to design a definitive large-scale clinical trial.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (intervention): Patients undergo a home-based, computerized, interactive training program comprising 3-5 sessions of 15-45 minutes every week for 5-9 weeks. The program contains twelve visually engaging and interesting exercises that target skills involving visual-spatial and verbal working memory (WM). The program is adaptive in a way that each difficulty task is automatically adjusted on a trial-by-trail basis to match a patient's current WM. Each patient has an interventional coach who has online access to patient's training sessions and outcomes (pass or fail). Coaches are able to modify the training sequence or make suggestions to patients and/or parents about how progress can be maximized. Coaches also have telephone meetings with patients and/or families once a week to ensure compliance, track progress, provide feedback, and answer questions that arise during training.

ARM II (control): Patients undergo a home-based, computerized, interactive, non-adaptive training program comprising 3-5 sessions of 15-45 minutes a week for 5-9 weeks. Each patient also has an interventional coach as in arm I. Patients in both arms complete a brief neuropsychological/behavioral assessment comprising the Wechsler Intelligence Scale for Children (WIS-IV), the Children's Memory Scale (CMS), and the California Verbal Learning Test-Children's Version (CVLT-C) at baseline, after completion of study, and at 6 months after completion of study. Additionally, parents complete a parent-report questionnaire to gather information about patient's behaviors, thoughts, emotions, adaptive skills, and social and functional impairment. Parents and children also complete surveys about the program regarding technical feasibility, adherence, ease-of-use, and satisfaction.

After completion of study treatment, participants are followed up within 3 weeks, then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be newly diagnosed or relapsed/progressed with a brain tumor that has not previously been treated with CRT

  * Note: COG therapeutic study participation is not required for ACCL10P1 enrollment
* Patient enrollment must occur within 4 calendar months following completion of CRT

  * Reminder: after patient enrollment, baseline testing followed by randomization must occur within 2-4 months after completion of CRT
* The patient must have an identified caregiver who is willing and able to oversee the training practice during the intervention period (ie, for 5-9 weeks starting approximately 3 months after completion of CRT)
* The patient must have access to a telephone and phone number where they can be reached
* The patient and caregiver must have reading, speaking and listening comprehension of English
* All patients and/or their parents or legal guardians must sign a written informed consent (patient assent is also recommended when applicable according to each institution's policy)
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with pontine glioma are not eligible
* Patients with an estimated survival of less than one year are not eligible
* Patients with a history of traumatic brain injury prior to tumor diagnosis are not eligible
* Patients with a motor, visual, or auditory handicap that prevents computer use (e.g., unresolved posterior fossa syndrome) are not eligible to participate in this trial
* Patients with full-scale intelligence quotient (IQ) < 70 per previous testing OR existing diagnosis of/educational classification as a student with an intellectual disability are not eligible

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina K Hardy, Principal Investigator — Children's Oncology Group
Locations (28):
- United States (27):
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Blank Children's Hospital, Des Moines, Iowa
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 45 total enrollments, among which 3 were never assigned to a treatment arm.
Groups:
- No Assigned Arm: Patients never assigned to a treatment arm.
Period: Overall Study
Arm/Group | Arm I (Interactive Training Program) | Arm II (Non-adaptive Training Program) | No Assigned Arm
Started | 21 | 21 | 3
Completed | 11 | 11 | 0
Not Completed | 10 | 10 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Did Not Start Treatment | 4 | 3 | 3
Not completed — Progressive disease | 3 | 1 | 0
Not completed — Patient did not complete cognitive training within 9 weeks | 3 | 3 | 0
Not completed — Refusal of further protocol therapy by patient/parent/guardian | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Interactive Training Program) | Arm II (Non-adaptive Training Program) | No Assigned Arm | Total
Number analyzed (Participants) | 21 | 21 | 3 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 3 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (2.7) | 10.6 (3) | 11.7 (2.9) | 10.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 1 | 15
  Male | 14 | 14 | 2 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 14 | 18 | 3 | 35
  Unknown or Not Reported | 5 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 1 | 4
  White | 11 | 17 | 2 | 30
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 5 | 1 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 4 | 0 | 9
  United States | 16 | 17 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: Intervention Compliance
Description: Intervention compliance is defined as at least 80% of computerized training sessions completed (i.e., completing at least 20 sessions within 9 weeks of starting training). Will report the proportion of eligible, randomized patients who meet the compliance definition by arm with corresponding 95% confidence intervals.
Time Frame: Up to 9 weeks of starting training
Population: Per protocol, the analysis includes all eligible, randomized participants without a medical event during cognitive training (cancer relapse/progression, death, removal from protocol therapy due to physician's determination in the patient's best interest, development of seizures or other change in functional status, or starting or changing the dose of psychostimulants).
  dose of psychostimulants)."
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Arm I (Interactive Training Program) | Arm II (Non-adaptive Training Program)
Number analyzed (Participants) | 18 | 20
Proportion of Participants | 0.39 [0.17 to 0.64] | 0.50 [0.27 to 0.73]

2. Other Pre Specified Outcome: Parent-rated Executive Function Using the Metacognition Subscales From the Behavior Rating Inventory of Executive Function (BRIEF)
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Working Memory (WM) Using the Metacognition Subscales From (BRIEF)
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Executive Function Using the Groton Maze Learning Task of the CogState Battery
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: WM by the One-back Task From CogState
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

6. Other Pre Specified Outcome: WM by Digit Span From Wechsler Intelligence Scales
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Visual Working Memory Using Spatial Span From Wechsler Scale
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Visual Memory Using Dot Location From Children's Memory Scale
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Technical Feasibility Based on the Item Responses to the 13-item Feasibility Interview
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Adherence Based on Total Number of Training Sessions Completed
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Satisfaction Based on the Item Responses to the 13-item Feasibility Interview
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Ease of Use Based on the Item Responses to the 13-item Feasibility Interview
Description: Descriptive/summary statistics will be provided.
Time Frame: Up to 6 months post training completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Arm I (Interactive Training Program) | Arm II (Non-adaptive Training Program) | No Assigned Arm
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT01503086/Prot_SAP_000.pdf